CLINICAL TRIAL: NCT01337323
Title: Prospective Observational Study of Concomitant Allergic Rhinitis Treatment Patterns Among Patients Starting on Fluticasone Furoate Nasal Spray in a Retail Pharmacy Setting
Status: Terminated | Type: Observational
Why Stopped: Insufficient number of patient records met inclusion criteria
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112602
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Rhinitis, Allergic, Seasonal; Seasonal Allergic Rhinitis
Keywords: allergic rhinitis, allergies, concomitant medications, allergy symptoms
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- New prescription for fluticasone furoate nasal spray: patients receiving their first prescription for fluticasone furoate nasal spray and who have active seasonal allergic rhinitis with a history of using another intranasal steriod (INS) and other concomitant allergic rhinitis medications to treat their seasonal allergy symptoms.
  Interventions: Drug: Fluticasone furoate nasal spray

INTERVENTIONS:
Drug: Fluticasone furoate nasal spray — fluticasone furorate intranasal steroid spray
  Other Names: Flonase® is a registered trademark of GlaxoSmithKline

SUMMARY:
This study is a prospective observational cohort study with 3-month follow-up among a cohort of intranasal steroid (INS) -experienced patients newly starting fluticasone furorate nasal spray (FFNS). The primary aim is to examine the effect of FFNS on the use and associated cost of concomitant allergic rhinitis medications in INS-experienced patients starting treatment with FFNS who have a history of prior concomitant medication use. The secondary aim will be to determine the effect of FFNS on control of allergic rhinitis, as assessed by the Rhinitis Control Assessment Test (RCAT).

Adult patients filling a new FFNS prescription will be recruited (within 4 days of starting their FFNS) across 50 branches of a retail pharmacy chain with co-located convenient care clinics. Approximately 350 patients who have active seasonal rhinitis and have used an INS other than FFNS and another prescription or over-the-counter allergy medication in the previous allergy season will be eligible for the study. A baseline questionnaire will be administered to collect information on patient demographics, a brief medical history of the patient's rhinitis, prior use of INS and other prescription and over-the-counter medications taken for allergic rhinitis, total out of pocket costs for the prior allergy season, number of office visits due to allergic rhinitis, and level of control of symptoms of allergic rhinitis.

At 1, 2, and 3 months post-enrollment, a follow-up questionnaire will be administered to collect information on medications taken for allergic rhinitis, office visits due to rhinitis, and level of control of symptoms of allergic rhinitis. In addition, pharmacy claims data will be abstracted for patients 1 year prior to enrollment and 4 months after enrollment to verify and supplement patient reported data as needed.

The primary outcomes will be rate of use of non-INS concomitant medications (frequency and duration) at baseline, and 1, 2, and 3 months follow-up and change in rate of use of non-INS concomitant medications (post vs. pre and from baseline to 3 months follow-up). Secondary outcomes will be change in total allergic rhinitis pharmacy expenditures (post vs. pre and from baseline to follow-up) and change in the level of control of allergic rhinitis, as measured by score on the Rhinitis Control Assessment Test (RCAT), from baseline to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Active seasonal allergic rhinitis
* Initiating first-time treatment with fluticasone furoate nasal spray (FFNS)
* Received treatment with at least one intra-nasal steroid (INS) other than FFNS during the last allergy season
* Received treatment with one or more antihistamines, leukotriene receptor atagonists (LTRA), topical ocular medications, or any over the counter (OTC) medication for allergic rhinitis symptoms during the last allergy season
* At least 18 years of age at the time of study enrollment
* Able to read, comprehend, and record information in English
* Have provided an appropriately signed and dated informed consent

Exclusion Criteria:

* Received prior treatment with FFNS
* Pregnant
* Employee or family members of an employee of the study sponsor, retail pharmacy chain, or convenient care clinic implementing the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients filling a new fluticasone furorate nasal spray (FFNS) prescription will be recruited across 50 branches of a retail pharmacy chain with co-located convenient care clinic located throughout the United States. Approximately 350 patients who have active seasonal rhinitis and have used an intra-nasal steroid (INS) other than FFNS and another prescription or over-the-counter allergy medication in the previous allergy season will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Non-intranasal steroid concomitant medication use | 3 months
  change in rate of non-intranasal steroid concomitant medication use (frequency and duration)

SECONDARY OUTCOMES:
Concomitant Medication Cost | 3 months
  Change in total allergic rhinitis pharmacy expenditures
RCAT Score | 3 months
  Level of control of allergic rhinitis, as measured by score on the Rhinitis Control Assessment Test (RCAT)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline